CLINICAL TRIAL: NCT03069118
Title: Effectiveness of a Remote Behavioral Intervention and Coaching Support for Risky Substance Users in a Randomized Control Trial
Brief Title: 90-Day Online Substance Use Program
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Workit Health (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: #2016/10/11
Record Dates: First submitted 2017-02-27; First posted 2017-03-03 (Actual); Last update posted 2017-03-13 (Actual); Status verified 2017-02

CONDITIONS: Addictive Behavior; Alcohol Use Disorder; Alcohol Abuse; Drug Abuse; Drug Use Disorders
Keywords: Telemedicine; Online Treatment; Digital Intervention
MeSH Terms: conditions — Behavior, Addictive; Alcoholism; Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental): Three-month intervention on the online Workit Health platform
  Interventions: Behavioral: Treatment - Workit Health Online Program
- Control (Placebo Comparator): A list of online resources/waitlist
  Interventions: Behavioral: Control - Resource List

INTERVENTIONS:
Behavioral: Treatment - Workit Health Online Program — The Workit Health program is an adaptive "recovery in your pocket" harm reduction and sobriety solution that provides 24-hour access to adaptive lessons, mentorship, written and audio driven therapeutic exercises and tools, and peer-to-peer coaching. Users access our online site and enter an initial 90-day program that takes a holistic approach to recovery by addressing the physical, mental, emotional, and social aspects of addiction. As they advance, they move through successive levels that include lessons, activities, and assignments. Bonus materials, such as meditations and suggested reading, give users timely opportunities to dive deeper into a problem they are struggling with that day. Workit Health implements evidence-based strategies such as CBT, DBT, and MI.
  Arms: Treatment
Behavioral: Control - Resource List — Tailored list of resources.
  Arms: Control

SUMMARY:
Individuals indicating risky substance use are randomly assigned either to a three-month online intervention on the Workit Health platform or a waitlist/treatment as usual. Those randomized to treatment will report reduced consumption of alcohol and other drugs and higher quality of life at study conclusion.

ELIGIBILITY:
Inclusion Criteria:

* Subjects of this research are adults who self-identify as wanting to change their relationship to alcohol or drugs, who report currently using alcohol or drugs, or having recently stopped, who have access to an internet-enabled device, who are not currently suffering from untreated acute medical or psychiatric conditions, who anticipate being able to access the intervention over a six-month period, and who are able to freely consent to participate by themselves.

Exclusion Criteria:

* Because the intervention is written for an adult audience, as well as the logistical challenges of having private access to an internet enabled device, this research is limited to participants over the age of 18.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2017-08-01 (Estimated); Study Completion 2017-12-01 (Estimated)

PRIMARY OUTCOMES:
ASSIST | 90-day
  The Alcohol, Smoking and Substance Involvement Screening Test
WHOQOL-BREF | 90-day
  World Health Organization Quality of Life (BREF) Questionnaire

SECONDARY OUTCOMES:
Net Promoter Score | 90-day
  User Satisfaction Survey

CONTACTS AND LOCATIONS:
Overall Officials: Lisa McLaughlin, Principal Investigator — Workit Health
Locations (1):
- Workit Health, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No